CLINICAL TRIAL: NCT04454099
Title: A Comparison of Quantitative Fecal Immunochemical Test and Qualitative Fecal Occult Blood Test for Colorectal Cancer Screening in Medium and High Risk Screening Population
Brief Title: A Comparison of Different Fecal Occult Blood Test for Colorectal Cancer Screening
Status: Completed | Type: Observational
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Clinical Professor, Shandong University
Other Study IDs: 2020SDU-QILU-524
Record Dates: First submitted 2020-06-09; First posted 2020-07-01 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; fecal occult blood testing; quantitative fecal immunochemical test
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fecal Occult Blood Test: People in this group will use four kind of fecal occult blood test, including quantitative and qualitative method, to detect Hb in stool before colonoscopy.
  Interventions: Diagnostic Test: 4 kind of FOBT and colonoscopy with pathological examination

INTERVENTIONS:
Diagnostic Test: 4 kind of FOBT and colonoscopy with pathological examination — Detect Hb in stool by 4 kind of FOBT and detect colon lesion using colonoscopy and pathological examination.

SUMMARY:
Colorectal cancer is a leading cause of cancer-related morbidity and mortality. CRC-related death can be prevented through fecal occult blood test screening. Because of economic and high sensitivity, fecal immunochemical test is recommended for screening population of CRC. The purpose of this study is to compare the accuracy of 4 different fecal occult blood testing in medium and high risk screening population in Chinese.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is one of the most common cancer worldwide, and cause a huge number of cancer-associated mortality. CRC screening has been shown to be effective in reducing the incidence of, and mortality from, CRC. There are several recommended screening options for screening population of CRC, including colonoscopy and fecal occult blood testing (FOBT) .Colonoscopy has higher sensitivity and specificity than FOBT for detecting advanced colorectal neoplasia but also has several disadvantages, including higher cost and poorer compliance. Therefore, many patients prefer FOBT to colonoscopy. FOBT includes guaiac-based fecal occult blood test (gFOBT) and fecal immunochemical test (FIT). FIT includes quantitative FIT (qFIT) and qualitative FIT. qFIT can provide a value of concentration of hemoglobin in stool and are increasingly recommended for CRC. In China, the most common use FOBT is qualitative FIT and the comparison of quantitative and qualitative FIT is lack in screening population of CRC in Chinese. To add to the evidence on FIT performance characteristics for detection of CRC, the investigators design this research to compare qFIT with other 3 qualitative FOBT（two of them are colloidal gold qualitative FITs and one of them is chemical and immunologic combined detection）in medium and high risk screening population.

ELIGIBILITY:
Inclusion Criteria:

* Adults 50-75 years old;
* Asia-Pacific Colorectal Screening score(APCS): medium or high risk.

Exclusion Criteria:

* APCS score: low risk;
* People with history of intestinal surgery;
* People with history of CRC;
* People with history of inflammatory bowel disease, ischemic enteritis, vascular malformation of intestine or other disease resulting in intestinal tract bleeding;
* People with symptoms including visible rectal bleeding, hematuria, severe and acute diarrhea and Bristol feces score 7th type;
* Pregnancy, lactation or menstrual phase;
* Severe congestive heart failure or other sever disease cause cannot tolerate colonoscopy.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Continuous participants intending to undergo colonoscopy and meet the inclusion and exclusion criteria from Qilu Hospital were enrolled.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-03-18 (Actual)

PRIMARY OUTCOMES:
The accuracy of 4 kind of FOBTs to diagnose CRC. | 6 months
  The sensitivity, specificity, positive predictive value and negative predictive value of these 4 FOBTs to detect CRC.
The accuracy of 4 kind of FOBTs to diagnose advanced colorectal neoplasm. | 6 months
  The sensitivity, specificity, positive predictive value and negative predictive value of these 4 FOBTs to detect advanced colorectal neoplasm.
The accuracy of 4 kind of FOBTs to diagnose advanced adenoma. | 6 months
  The sensitivity, specificity, positive predictive value and negative predictive value of these 4 FOBTs to detect advanced adenoma.
Develop a predictive model of CRC or advanced colorectal neoplasm which includes qFIT. | 6 months
  Develop a predictive model of CRC or advanced colorectal neoplasm which includes qFIT, age ,sex, CRC family history and so on.

SECONDARY OUTCOMES:
Explore the cost-benefit ratio of one or two-sample of qFIT. | 6 month
  Explore the cost-benefit ratio of one or two-sample of qFIT.
Explore the reason of false positive of qFIT | 6 month
  Calculate false positive rate of the 4 kind of FOBTs. and count the case number of inflammatory bowel disease, colonic diverticulitis, hemorrhoids, upper gastrointestinal disease or medical factors that cause false positive of qFIT.
Explore the effect of aspirin or other anticoagulants to the diagnose accuracy of qFIT | 6 month
  Count sensitivity and specificity with or without patients who take aspirin or other anticoagulants.

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, PhD, Study Chair — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Robertson DJ, Lee JK, Boland CR, Dominitz JA, Giardiello FM, Johnson DA, Kaltenbach T, Lieberman D, Levin TR, Rex DK. Recommendations on Fecal Immunochemical Testing to Screen for Colorectal Neoplasia: A Consensus Statement by the US Multi-Society Task Force on Colorectal Cancer. Gastroenterology. 2017 Apr;152(5):1217-1237.e3. doi: 10.1053/j.gastro.2016.08.053. Epub 2016 Oct 19. PMID 27769517